CLINICAL TRIAL: NCT03936686
Title: Assessment of the Knowledge Level Regarding Cardiovascular Disease Risk Factors: Comparison Across Age Groups
Brief Title: CVD Risk Factor Knowledge Across Age Groups
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: D'Youville College (Other)
Responsible Party: Principal Investigator, Pamela Bartlo, Clinical Associate Professor, D'Youville College
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CVD Risk Factor Knowledge
Record Dates: First submitted 2019-04-30; First posted 2019-05-03 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Cardiovascular Risk Factor
Keywords: Education; Knowledge level

STUDY DESIGN:
Intervention Model Description: There were five participant groups evaluated based on age groupings. These groups were compared within group and against each other.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Children in grades 4 or 5 (Active Comparator): This group was comprised of participants that were in grades 4 or 5 in school.
  Interventions: Other: Survey tool to assess CVD risk factor knowledge
- Adolescents in grades 10 or 11 (Active Comparator): This group was comprised of participants that were in grades 10 or 11 in school.
  Interventions: Other: Survey tool to assess CVD risk factor knowledge
- College Age Participants (Active Comparator): This group was comprised of participants that were sophomores or juniors in college/university that were non-health career majors.
  Interventions: Other: Survey tool to assess CVD risk factor knowledge
- Cardiac Rehab Adults (Active Comparator): This group was comprised of participants that were adults over the age of 40 that had completed a phase II cardiac rehabilitation program.
  Interventions: Other: Survey tool to assess CVD risk factor knowledge
- General Adults (Active Comparator): This group was comprised of participants that were adults over the age of 40 that had never attended an outpatient cardiac rehabilitation program before.
  Interventions: Other: Survey tool to assess CVD risk factor knowledge

INTERVENTIONS:
Other: Survey tool to assess CVD risk factor knowledge — The survey tool was used to assess the participant's knowledge level and their previous methods of education regarding cardiovascular disease risk factors.

SUMMARY:
This study was to examine the knowledge level regarding cardiovascular disease risk factors among participants of varying ages. Then to see if there was any type of previous education that led to greater knowledge levels.

DETAILED DESCRIPTION:
This study used a survey tool that assessed the participants' method(s) of prior education regarding cardiovascular disease (CVD) risk factors. Then the participant was asked eleven questions regarding CVD risk factors which tested their knowledge of those factors. Analysis was done to evaluate overall knowledge level of each group and compare the knowledge levels across age groups. Then analysis was done to see if any method(s) led to better knowledge level within and/or between age groups.

ELIGIBILITY:
Inclusion Criteria:

* were specific to age for each participant group and then also included full completion of the survey for all groups.

Exclusion Criteria:

* age outside of specified population for each participant groups or incomplete survey for any participant regardless of group.

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 381 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Cardiovascular disease risk factor knowledge | 10-15 minutes
  How well did the participant know the risk factors for cardiovascular disease. This was determined by using a survey tool that was shown to have internal validity using Chronbach alpha score. The survey had 11 questions regarding CVD risk factors and asked the participant if they felt the statement was completely true, somewhat true, neutral, somewhat untrue, or completely untrue. Survey scores were determined out of 55 total points.
Method(s) of education | 10-15 minutes
  What methods of education regarding CVD risk factors did the participant previously have. The participant was asked various methods of previous education. These included school for younger participants, cardiac rehab for that group, TV, media, Internet, community groups, health care provider, family member experience, or family member discussion. The were tabulated individually and then comparisons were made within and between groups for methods of education used. Then these were correlated to survey scores too. These comparisons were made with chi-square with post-hoc tests, MANOVAs, and unpaired t-tests.

IPD SHARING:
Plan to Share IPD: Undecided
If other researchers would like to use data, non-identified results could be shared. Individual participant surveys would not be shared.

REFERENCES:
- [Derived] Bartlo P, Irion G, Voorhees J. Assessment of the Knowledge Level Regarding Cardiovascular Disease Risk Factors: Comparison Across Age Groups. J Community Health. 2020 Oct;45(5):1030-1037. doi: 10.1007/s10900-020-00824-w. PMID 32323174